CLINICAL TRIAL: NCT07334106
Title: Emotional Well-being and Biomarkers of Healthy Aging
Brief Title: Emotional Well-being and Measures of Healthy Aging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Potocsnak Human Longevity Lab (Unknown)
Responsible Party: Principal Investigator, Judith Moskowitz, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STU00221612
Record Dates: First submitted 2025-12-08; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Aging; Aging, Healthy; Aging Well; Aging, Biological
Keywords: Aging; Resilience, Psychological; Psychological Well-Being; Aging Well; Internet-Based Intervention
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This study is a waitlist-control design. Participants in the control participant will receive the positive psychology intervention at the conclusion of the study.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Emotion Skills Intervention (Experimental): Participants will receive the 6-week online intervention, PARK (Positive Affect Regulation sKills Course).
  Interventions: Behavioral: Positive Emotion Skills Intervention
- Waitlist Control (No Intervention): The waitlist control condition will receive usual care in the Human Longevity Lab, which consists of a feedback report on biological age and lifestyle counseling from a clinical provider at the end of the study period. Control condition participants will have the option to gain access to the PARK platform and learn positive emotion skills after their study participation is completed at the end of 12 months.

INTERVENTIONS:
Behavioral: Positive Emotion Skills Intervention — Skills include positive events, capitalizing, gratitude, mindfulness, positive reappraisal, personal strengths, achievable goals, and self-compassion. The skills will be delivered over approximately 6 weeks, and individuals can participate from any device and location with internet access. A week will consist of 1-2 days of didactic material and 5-6 days of real-life skills practice and reporting. Participants cannot skip ahead and can only progress to the next lesson if they have completed the current one, but they can return to old lessons or exercises if they wish to.
  Arms: Positive Emotion Skills Intervention

SUMMARY:
This randomized control study is designed to understand the role of a positive psychology intervention (PARK: Positive Affect Regulation sKills) in biological aging and well-being. PARK provides a series of positive emotion skills in a self-guided online format, making the program accessible and convenient.

Our main aims are:

Aim 1: To explore the effects of PARK on psychological well-being (e.g., depression, anxiety, positive affect).

Aim 2: To explore the effects of PARK on biological age as defined by DNA methylation (DNAm) GrimAge and electrocardiogram-age (ECG-age), as well as physiological well-being in adults (e.g., cardiovascular, endocrine, musculoskeletal functioning, etc.).

DETAILED DESCRIPTION:
The skills in the Positive Psychology Intervention (PPI), PARK (e.g., gratitude, mindful awareness and nonjudgement, and self-compassion) are designed to promote positive emotion, which has been shown to provide resilience against stress. Positive emotion, independent of stress and negative emotion, has also been associated with a lower risk of mortality and better health behaviors such as likelihood of physical activity and healthy eating. This randomized control study will compare baseline well-being scores to post-online intervention at 3 months, 6 months, and 12 months post-baseline. Secondarily, measures of biological aging (DNAm GrimAge and ECG-age) and physiological functioning measures of cardiovascular, musculoskeletal, and endocrine functioning will be explored from baseline to post-intervention measures 3 and 12 months later.

Research will be based in Northwestern's Feinberg School of Medicine through the Potocsnak Human Longevity Lab and the Department of Medical Social Sciences (MSS), with all study procedures conducted in-person at the Human Longevity Lab or online. Eligibility screening, consent, and assessments will be conducted on REDCap. Consenting participants randomized to the treatment group will receive access to the online PARK platform within two weeks. The intervention consists of a positive skills course (including weekly lessons and daily skills practice) and daily emotion check-ins, hosted by BrightOutcome. The skills will be delivered over approximately 6 weeks, and individuals can participate from any device and location with internet access.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70
* Speaks and reads English
* Able to access the online platform through their phone, a public device (i.e., at the library) or at home.
* Lives in the Chicagoland area
* Willing/able to travel to the Human Longevity Lab for in-person visits

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Vulnerable Populations
* Pre-existing heart disease (prevalent coronary heart and cerebrovascular disease or heart failure)
* Type 2 diabetes
* Severe psychiatric illness

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS) Positive Affect (v1.0) and PROMIS Meaning and Purpose (v1.0) | Baseline, 3 months, 6 months, 12 months
  Computer Adaptive Testing measure of positive emotion and purpose. Higher scores mean a better outcome (i.e., more positive emotion). Scores can range from 9-85, and a t-score of 50 represents the mean score for the United States general population with a standard deviation of 10.
PROMIS Depression (v1.0), Anxiety (v1.0), Social Isolation (v2.0) | baseline and 3, 6, 12 months post-baseline
  Computer Adaptive Testing measures of psychosocial well-being.
  Higher scores mean a worse outcome (i.e., more anxiety or depression). Scores can range from 9-85, and a t-score of 50 represents the mean score for the United States general population with a standard deviation of 10.

SECONDARY OUTCOMES:
Biological Age: DNA methylation GrimAge | Baseline, 3 months, 12 months
  Biological age as defined by DNA methylation GrimAge, an estimation of biological age in units of years.
ECG-age (electrocardiogram-age) | Baseline, 3 months, 12 months
  Artificial intelligence algorithm using electrocardiogram data to estimate participant's age in unit of years. Higher ECG-age equates to greater cardiovascular aging.
Telomere Length | Baseline, 3 months, 12 months
  Telomere length measures cellular aging, measured in kilobases (kb). Longer telomere length indicates less cellular aging (a better outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Potocsnak Human Longevity Lab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pressman SD, Cohen S. Does positive affect influence health? Psychol Bull. 2005 Nov;131(6):925-971. doi: 10.1037/0033-2909.131.6.925. PMID 16351329
- [Background] Moskowitz JT, Carrico AW, Duncan LG, Cohn MA, Cheung EO, Batchelder A, Martinez L, Segawa E, Acree M, Folkman S. Randomized controlled trial of a positive affect intervention for people newly diagnosed with HIV. J Consult Clin Psychol. 2017 May;85(5):409-423. doi: 10.1037/ccp0000188. Epub 2017 Mar 23. PMID 28333512
- [Background] Pressman SD, Jenkins BN, Moskowitz JT. Positive Affect and Health: What Do We Know and Where Next Should We Go? Annu Rev Psychol. 2019 Jan 4;70:627-650. doi: 10.1146/annurev-psych-010418-102955. Epub 2018 Sep 27. PMID 30260746
- [Background] Steptoe A, Wardle J. Positive affect measured using ecological momentary assessment and survival in older men and women. Proc Natl Acad Sci U S A. 2011 Nov 8;108(45):18244-8. doi: 10.1073/pnas.1110892108. Epub 2011 Oct 31. PMID 22042845
- [Background] Behr LC, Simm A, Kluttig A, Grosskopf Grosskopf A. 60 years of healthy aging: On definitions, biomarkers, scores and challenges. Ageing Res Rev. 2023 Jul;88:101934. doi: 10.1016/j.arr.2023.101934. Epub 2023 Apr 13. PMID 37059401
- [Background] Prior A, Fenger-Gron M, Larsen KK, Larsen FB, Robinson KM, Nielsen MG, Christensen KS, Mercer SW, Vestergaard M. The Association Between Perceived Stress and Mortality Among People With Multimorbidity: A Prospective Population-Based Cohort Study. Am J Epidemiol. 2016 Aug 1;184(3):199-210. doi: 10.1093/aje/kwv324. Epub 2016 Jul 11. PMID 27407085
- [Background] Yegorov YE, Poznyak AV, Nikiforov NG, Sobenin IA, Orekhov AN. The Link between Chronic Stress and Accelerated Aging. Biomedicines. 2020 Jul 7;8(7):198. doi: 10.3390/biomedicines8070198. PMID 32645916